CLINICAL TRIAL: NCT00275496
Title: A Clinical Study of Wide Excision Alone Versus Wide Excision With Intraoperative Lymphatic Mapping and Selective Lymph Node Dissection in the Treatment of Patients With Cutaneous Invasive Melanoma.
Brief Title: Multicenter Selective Lymphadenectomy Trial (MSLT)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Saint John's Cancer Institute (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MSLT-1; NIH P01 CA029605
Record Dates: First submitted 2006-01-10; First posted 2006-01-12 (Estimated); Last update posted 2015-09-02 (Estimated); Status verified 2014-05

CONDITIONS: Melanoma
Keywords: SLND; Sentinel; Melanoma; Surgical
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- WEX only (Active Comparator)
  Interventions: Procedure: Wide Excision
- WEX + SLND (Active Comparator)
  Interventions: Procedure: Sentinel Lymph Node Dissection
- WEX+SLND+CLND (Active Comparator)
  Interventions: Procedure: Complete Lymph Node Dissection

INTERVENTIONS:
Procedure: Sentinel Lymph Node Dissection — Subject has wide excision and sentinel lymph node dissection for primary melanoma.
  Arms: WEX + SLND
Procedure: Complete Lymph Node Dissection — Subject has wide excision, sentinel lymph node dissection, and complete lymph node dissection (if positive sentinel node found) for primary melanoma.
  Arms: WEX+SLND+CLND
Procedure: Wide Excision — Subject has wide excision only for primary melanoma.
  Arms: WEX only

SUMMARY:
Subjects must be diagnosed with melanoma. All subjects receive Wide Excision (WEX) of their melanoma. If the melanoma meets study requirements, the subject is randomized to receive either (1) no further surgical procedures as part of the study or (2) a Selective Lymphadenectomy with the possibility of a Complete Lymphadenectomy. Subjects are then followed for 10 years.

ELIGIBILITY:
Inclusion Criteria:

1. The patient consents to be in the study.
2. The patient must have invasive melanoma with: 1) Clark Level III and Breslow Thickness greater than or equal to 1.00 mm; or 2) Clark Level IV or V with any Breslow thickness. A confirmation of diagnosis and thickness must be made by the institutional pathologist.
3. The primary cutaneous melanoma site must be on the head, neck, trunk, extremity, scalp, palm of the hand, sole of the foot, or subungual skin.
4. The patient's biopsy must have been completed no more than 10 weeks before the initial visit to the clinic. (Surgery must be scheduled within three months of the biopsy.)
5. The patient must be between 18 and 75 years old.
6. The patient must have a life expectancy of at least 10 years from the time of diagnosis, excluding the diagnosis of melanoma.

Exclusion Criteria:

1. The patient had a prior wide excision of the primary with a diameter of excision greater than or equal to 3.0 cm and the shortest margin from the tumor edge to the excision edge was measured by a pathologist to be greater than or equal to 1.5 cm; or the patient had an elliptical excision and a margin beyond the tumor edge was greater than or equal to 1.5 cm at the narrowest margin.
2. The primary cutaneous melanoma involves the eye, ear, mucous membranes.
3. The patient has clinical evidence of satellite lesions, in-transit, regional nodal or distant metastases.
4. The patient has a second primary invasive melanoma.
5. The patient has had any type of solid tumor or hematologic malignancy during the past 5 years. Exceptions are if the patient has been treated for T1 lesions (e.g., squamous cell carcinoma of the skin, basal cell carcinoma or in situ carcinoma of the uterine cervix) during the past 5 years, but has not received treatment within the last 6 months.
6. The patient has had prior skin grafts, tissue transfers or flaps, or lymph node dissections that may alter the lymphatic drainage pattern from a primary cutaneous melanoma to the adjacent regional lymph node basins.
7. The patient has had previous chemotherapy, immunotherapy or radiation therapy.
8. The patient has had an organ transplantation and is receiving immunosuppressive agents as a result of the transplantation.
9. The patient has taken oral or parenteral steroids or immunosuppressive drugs within the last 6 months.
10. The patient has any known primary or secondary immune deficiencies.
11. The patient has another medical condition that will affect life expectancy.
12. The patient is pregnant.
13. Evidence that the patient cannot undergo selective lymph node dissection for any reason.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2001 (Actual)
Dates: Start 1993-11; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
To determine whether wide excision of the primary with intraoperative lymphatic mapping (LM) followed by selective lymphadenectomy will effectively prolong overall survival compared to wide excision of the primary melanoma alone. | 10 years

SECONDARY OUTCOMES:
Disease-free survival; Incidence, timing, and anatomic distribution of distant metastases; Morbidity of procedures; Significance of TA90 levels; Incidence of Sentinel Node Metastases (biopsy) vs clinical metastases (observation); Accuracy of LM | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Donald L Morton, MD, Study Chair — Saint John's Cancer Institute

REFERENCES:
- [Result] Morton DL, Thompson JF, Cochran AJ, Mozzillo N, Elashoff R, Essner R, Nieweg OE, Roses DF, Hoekstra HJ, Karakousis CP, Reintgen DS, Coventry BJ, Glass EC, Wang HJ; MSLT Group. Sentinel-node biopsy or nodal observation in melanoma. N Engl J Med. 2006 Sep 28;355(13):1307-17. doi: 10.1056/NEJMoa060992. PMID 17005948
- [Result] Faries MB, Thompson JF, Cochran A, Elashoff R, Glass EC, Mozzillo N, Nieweg OE, Roses DF, Hoekstra HJ, Karakousis CP, Reintgen DS, Coventry BJ, Wang HJ, Morton DL; MSLT Cooperative Group. The impact on morbidity and length of stay of early versus delayed complete lymphadenectomy in melanoma: results of the Multicenter Selective Lymphadenectomy Trial (I). Ann Surg Oncol. 2010 Dec;17(12):3324-9. doi: 10.1245/s10434-010-1203-0. Epub 2010 Jul 8. PMID 20614193
- [Result] Howard JH, Thompson JF, Mozzillo N, Nieweg OE, Hoekstra HJ, Roses DF, Sondak VK, Reintgen DS, Kashani-Sabet M, Karakousis CP, Coventry BJ, Kraybill WG, Smithers BM, Elashoff R, Stern SL, Cochran AJ, Faries MB, Morton DL. Metastasectomy for distant metastatic melanoma: analysis of data from the first Multicenter Selective Lymphadenectomy Trial (MSLT-I). Ann Surg Oncol. 2012 Aug;19(8):2547-55. doi: 10.1245/s10434-012-2398-z. Epub 2012 May 31. PMID 22648554
- [Derived] Morton DL, Thompson JF, Cochran AJ, Mozzillo N, Nieweg OE, Roses DF, Hoekstra HJ, Karakousis CP, Puleo CA, Coventry BJ, Kashani-Sabet M, Smithers BM, Paul E, Kraybill WG, McKinnon JG, Wang HJ, Elashoff R, Faries MB; MSLT Group. Final trial report of sentinel-node biopsy versus nodal observation in melanoma. N Engl J Med. 2014 Feb 13;370(7):599-609. doi: 10.1056/NEJMoa1310460. PMID 24521106